CLINICAL TRIAL: NCT07096362
Title: A Phase 2 Study Assessing Utility of ctDNA in Early Switch of First-line mFOLFIRINOX in Metastatic Pancreatic Ductal Adenocarcinoma
Brief Title: Utility of ctDNA in Early Switch of First-line mFOLFIRINOX in Metastatic Pancreatic Ductal Adenocarcinoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Miami (Other)
Collaborators: National Cancer Institute (NCI) (NIH); BillionToOne, Inc (Unknown)
Responsible Party: Principal Investigator, Gretel Terrero, Professor, University of Miami
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 20250087; K12CA226330 (NIH); NCI-2025-06277 (Registry Identifier: NCI Clinical Trials Reporting Program (NCI CTRP))
Record Dates: First submitted 2025-07-24; First posted 2025-07-31 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Metastatic Pancreatic Ductal Adenocarcinoma; Pancreatic Ductal Adenocarcinoma
MeSH Terms: interventions — Fluorouracil; Oxaliplatin; Leucovorin; Irinotecan; Gemcitabine; Taxes

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Part 1: Early Switch of Chemotherapy Interventional Cohort (Experimental): Participants in this group will receive ctDNA monitoring in combination with standard of care (SOC) of 5-fluorouracil, leucovorin, irinotecan, oxaliplatin (mFOLFIRINOX). Participants will receive standard of care treatment for up to 8 months.
  Total participation duration is approximately 18 months.
  Interventions: Drug: 5-Fluorouracil; Drug: Oxaliplatin; Drug: Leucovorin; Drug: Irinotecan; Diagnostic Test: Circulating Tumor Deoxyribonucleic acid (ctDNA) Assay
- Part 2 Arm A: Early Switch of Chemotherapy Interventional Cohort (Active Comparator): Participants in this group will receive ctDNA monitoring in combination with standard of care (SOC) of 5-fluorouracil, leucovorin, irinotecan, oxaliplatin (mFOLFIRINOX). After completing three cycles of therapy, participants with methylated-ctDNA fold change of less than threshold determined in Part 1 will continue to receive additional cycles of mFOLFIRINOX for up to 8 months. Participants with methylated-ctDNA fold-change of greater than threshold determined in Part 1 may switch to Part 2 Arm B.
  Total participation duration is approximately 18 months.
  Interventions: Drug: 5-Fluorouracil; Drug: Oxaliplatin; Drug: Leucovorin; Drug: Irinotecan; Diagnostic Test: Circulating Tumor Deoxyribonucleic acid (ctDNA) Assay
- Part 2 Arm B: Early Switch of Chemotherapy Interventional Cohort (Experimental): Participants in this group will receive ctDNA monitoring in combination with standard of care Gemcitabine and Nab-Paclitaxel therapy, after completion of up to three cycles of mFOLFIRINOX from Part 2 Arm A. Participants will receive standard of care treatment for up to 8 months.
  Total participation duration is approximately 18 months.
  Interventions: Drug: 5-Fluorouracil; Drug: Oxaliplatin; Drug: Leucovorin; Drug: Irinotecan; Drug: Gemcitabine; Drug: Nab Paclitaxel; Diagnostic Test: Circulating Tumor Deoxyribonucleic acid (ctDNA) Assay

INTERVENTIONS:
Drug: 5-Fluorouracil — Participants will be administered 2400 mg/m^2 of 5-Fluorouracil via continuous intravenous infusion over a 46-hour period beginning on Day 1 of each two-week cycle of standard of care (SOC) modified Folfirinox combination therapy.
Drug: Oxaliplatin — Participants will be administered 85 mg/m^2 of Oxaliplatin via intravenous infusion beginning on Day 1 of each two-week cycle of standard of care (SOC) modified Folfirinox combination therapy.
Drug: Leucovorin — Participants will be administered 400 mg/m^2 of Leucovorin via intravenous infusion beginning on Day 1 of each two-week cycle of standard of care (SOC) modified Folfirinox combination therapy.
Drug: Irinotecan — Participants will be administered 150 mg/m^2 of Irinotecan via intravenous infusion beginning on Day 1 of each two-week cycle of standard of care (SOC) modified Folfirinox combination therapy.
Drug: Gemcitabine — Participants will be administered 1000 mg/m^2 of Gemcitabine standard of care (SOC) via intravenous infusion on days 1, 8 and 15 of each four-week treatment cycle.
  Arms: Part 2 Arm B: Early Switch of Chemotherapy Interventional Cohort
Drug: Nab Paclitaxel — Participants will be administered 125 mg/m^2 of Nab Paclitaxel standard of care (SOC) by intravenous infusion on days 1, 8 and 15 of each four-week treatment cycle.
  Arms: Part 2 Arm B: Early Switch of Chemotherapy Interventional Cohort
Diagnostic Test: Circulating Tumor Deoxyribonucleic acid (ctDNA) Assay — ctDNA will be measured in participants in person via blood samples during Screening/Baseline and at the following intervals during treatment and follow-up:
  * Every weeks 2 beginning at weeks 2, 4, 6 and 8 of standard of care therapy.
  * Every 4 weeks beginning at week 10 of standard of care therapy until disease progression.
  ctDNA will be measured to obtain participant tumor methylation scores (TMS).

SUMMARY:
The purpose of this study is to understand whether a blood-based test called circulating tumor DNA (ctDNA) can detect whether participants are having a desired tumor shrinkage or an undesired lack of tumor shrinkage, and to study whether these levels of ctDNA can be used to make treatment decisions faster than the current standard approach, which is to wait 8 weeks after starting chemotherapy to obtain participant first imaging scans since starting chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed, metastatic pancreatic adenocarcinoma. Patients with adenosquamous carcinoma and mixed adenocarcinoma/neuroendocrine carcinoma (MANEC) of the pancreas are eligible, but pure neuroendocrine neoplasms are excluded.
2. Treatment-naïve patients diagnosed with metastatic pancreatic adenocarcinoma.
3. Must have a detectable circulating tumor deoxyribonucleic acid (DNA) at cycle 1 day 1.
4. Patients must have a detectable circulating tumor deoxyribonucleic acid (ctDNA) quantity on Northstar Response assay at baseline.
5. At least one tumor measurable by Computed Tomography (CT) scan or Positron Emission Tomography-Computed Tomography (PET/CT) scan. Measurable disease is defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded for non-nodal lesions and short axis for nodal lesions) as >20 mm with conventional techniques or >10 mm with spiral CT scan.
6. Adult male and female participants (≥ 18 years of age).
7. Male or non-pregnant and non-lactating female. Men and women with intact reproductive potential must agree to use contraception.
8. Adequate biological parameters as demonstrated by the following blood counts at Screening (obtained ≤ 21 days prior to enrollment) and at Baseline-Day 0:

   * Absolute neutrophil count (ANC) ≥ 1.0 × 109 cells/L.
   * Platelet count ≥ 100,000 cells/mm3 (100 × 109 cells/L). Supportive platelet transfusions are acceptable.
   * Hemoglobin (Hgb) ≥ 9 g/dL. Supportive packed red blood cell transfusions are acceptable.
9. Adequate blood chemistry levels at Screening (obtained ≤ 21 days prior to enrollment) and at Baseline-Day 0:

   * Aspartate aminotransferase (AST) - serum glutamic-oxaloacetic transaminase (SGOT); alanine transaminase (ALT) - serum glutamic-pyruvic transaminase (SGPT) ≤ 2.5 × upper limit of normal (ULN) range, unless liver metastases are present, then ≤ 5 × ULN is allowed.
   * Total bilirubin ≤ 1.5 × Upper Limit of Normal.
   * Estimated creatinine clearance of > 60 mL/min (per Cockcroft-Gault formula).
   * Albumin ≥ 3.0 g/dL.
10. Eastern Cooperative Oncology Group (ECOG) performance status from 0 to ≤ 1.
11. Must be a modified Folfirinox chemotherapy candidate.
12. For participants not qualified or able to give legal consent, consent must be obtained from their legally authorized representative (LAR).

Exclusion Criteria:

1. Patients with pure neuroendocrine neoplasms of the pancreas.
2. Brain metastases.
3. Uncontrolled ascites.
4. Increase of ECOG to > 1 between screening and enrollment.
5. Active, uncontrolled bacterial, viral, or fungal infection(s) requiring systemic therapy.
6. History of untreated or uncontrolled HIV and/or Hepatitis B or C infection.
7. Clinically significant, uncontrolled heart disease and/or cardiac repolarization abnormality, including any of the following:

   * History of myocardial infarction, angina pectoris, symptomatic pericarditis, or coronary artery bypass graft within six months prior to study entry
   * Documented cardiomyopathy
8. Grade 2 or greater sensory peripheral neuropathy.
9. History of chronic diarrhea.
10. Pregnant or nursing.
11. Concomitant serious medical or psychiatric illness that, in the opinion of the investigator, could compromise the patient's safety or integrity of the study data.
12. Concurrently enrolled in any other interventional clinical protocol or investigational trial involving administration of antineoplastic compounds for the treatment of metastatic pancreatic cancer.
13. Patient is unwilling or unable to comply with study procedures.
14. Patients with impaired decision-making capacity.
15. No other medical condition or reason that, in the opinion of the investigator, would preclude study participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-09-09 (Actual); Primary Completion 2030-09-30 (Estimated); Study Completion 2030-09-30 (Estimated)

PRIMARY OUTCOMES:
Part 1:Change in ctDNA fold-change at Week 4 | Baseline, Up to 4 weeks (after intervention)
  Circulating tumor Deoxyribonucleic Acid (ctDNA) fold-change at week 4 is defined as the ratio between ctDNA quantity at week 4 relative to baseline. The quantity of ctDNA will be measured in ng/mL.
  At week 4 among participants in Part 1 will be reported as a Tumor Methylation Score (TMS) in plasma samples. The ratio between the TMS at week 4 (TMS4) and the TMS at baseline (TMS0) will be calculated.
Part 1: Number of Radiographic Response Status Responders vs. Number of Non-Responders | Up to 1.5 years (after intervention)
  Radiographic response status among participants in Part 1 will be reported in numbers. Participants will undergo Positron Emission Tomography/Computed Tomography (PET/CT) radiographic imaging scans at the end of week 8. Participants will be subdivided into two groups: responders vs. non-responders to modified Folfirinox treatment. Responders will be defined as the number of participants achieving complete response (CR), partial response (PR) or exhibiting stable disease (SD). Non-responders will be defined as the number of participants exhibiting progressive disease (PD). Response will be evaluated using Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 criteria.
Part 2: Progression-Free Survival (PFS) | Up to 3.5 years (after intervention)
  Progression-Free Survival (PFS) is defined as elapsed time in months from day 1 of starting second-line (2L) chemotherapy until the date of documented progressive disease (PD) or death.

SECONDARY OUTCOMES:
Part 1: Change in ctDNA Tumor Methylation Score (TMS) | Baseline, Up to 8 weeks (after intervention)
  Circulating tumor Deoxyribonucleic Acid (ctDNA) Tumor Methylation Score (TMS) is defined as the amount of methylated tumor DNA in the blood. ctDNA TMS will be assessed at baseline, weeks 2, 4, 6, and 8.
  The Tumor Methylation Score (TMS) score ranges from 10 to 1,000,000. TMS is proprietary score, it does not have units. Higher TMS means higher levels of methylated tumor DNA found in the blood.
Part 1: Number of Radiographic Responses | Up to 8 weeks (after intervention)
  The number of radiographic response among participants in Part 2 will be reported as the result of Positron Emission Tomography/Computed Tomography (PET/CT) radiographic imaging scans taken at the end of week 8. Response will be evaluated using Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 criteria.
Part 2: Overall Survival (OS) | Up to 3.5 years (after intervention)
  Overall Survival (OS) is defined as elapsed time in months from start of first-line (1L) mFOLFIRINOX treatment to date of death.

CONTACTS AND LOCATIONS:
Overall Officials: Gretel Terrero, MD, Principal Investigator — University of Miami
Locations (1):
- University of Miami, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No